CLINICAL TRIAL: NCT01269112
Title: Citrate-based Regional Anticoagulation Versus Heparin for Continuous Renal Replacement Therapy in Critically Ill Patients With Acute Renal Failure: a Randomized Controlled Trial
Brief Title: Citrate-based Regional Anticoagulation Versus Heparin for Continuous Renal Replacement Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Patrick Saudan, PD Dr Patrick Saudan, MD, University Hospital, Geneva
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-069(NAC 09-27)
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2016-05

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- heparin (Placebo Comparator): CVVHDF performed using unfractionated heparin as anticoagulant and Prismasol as reinjection and dialysate fluids
  Interventions: Device: citrate regional anticoagulation
- citrate regional anticoagulation (Active Comparator): CVVHDF performed using Prismocitrate 18/0 solution (Trisodium citrate 18 mmol/L
  Interventions: Device: citrate regional anticoagulation

INTERVENTIONS:
Device: citrate regional anticoagulation — Patients randomly allocated to 2 treatment groups:
  Treatment A: - Regional citrate-based anticoagulation with the Prismocitrate® 10/2 solution (GAMBRO) Treatment B: - Standard unfractionated heparin anticoagulation
  Arms: heparin
Device: citrate regional anticoagulation — Patients randomly allocated to 2 treatment groups:
  Treatment A: - Regional citrate-based anticoagulation with the Prismocitrate® 10/2 solution (GAMBRO) Treatment B: - Standard unfractionated heparin anticoagulation

SUMMARY:
Critically ill patients with acute kidney injury (AKI) are at high risk of bleeding on account of coagulopathy, platelet dysfunction, frequent liver dysfunction and invasive procedures.In patients at high risk of bleeding, anticoagulation restricted to the circuit (regional anticoagulation) has been advocated as the method of choice.However, citrate anticoagulation may have many metabolic consequences, such as metabolic alkalosis due to citrate metabolism into bicarbonate, and in patients with liver disease, metabolic acidosis and hypocalcemia may occur.Implementation of citrate-based regional anticoagulation with frequent monitoring of acid-base and electolytes is also more challenging for the nurses and does not eliminate the need of a low-dose systemic anticoagulation for thromboses prophylaxis in most of the patients. Citrate-based regional anticoagulation is therefore mainly advocated only for patients at high-risk of bleeding.

The investigators plan to implement an open-label randomized control trial assessing the effectiveness of citrate-based regional anticoagulation in critically ill patients with AKI and with a special emphasis on the safety profile of this treatment in patients with severe liver failure.

DETAILED DESCRIPTION:
monocentric prospective open-label randomized controlled trial at the ICU of the University Hospitals of Geneva (Switzerland).

ICU patients eligible if they 18 yr old and had an AKI requiring CRRT Exclusion criteria Patients excluded if they had active hemorrhagic disorders or severe thrombocytopenia (< 50x109/L), a history of heparin-induced thrombocytopenia, severe liver failure defined as a factor V <20% or were on the waiting list for liver transplantation.

Treatment assignment Subjects enrolled into the trial randomly allocated to either heparin or citrate anticoagulation

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute kidney injury requiring renal replacement therapy (RIFLE criteria)
* Patients (males or females) > 18 yrs old
* Consent form signed (or in emergency investigator's statement form)

Exclusion Criteria:

* Patients with active bleeding disorders
* Patients with past history of heparin-induced thrombocytopenia (HIT)
* Patients with very severe liver disease ( patients awaiting liver transplant or factor V < 20% or MELD score > 25)
* Pregnancy (negative pregnancy test required in child-bearing age women prior to inclusion)
* Enrollment in another concurrent therapeutic trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-11; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Mean daily dialysis delivered dose during intensive care stay | dialysis days during intensive care stay
  * Mean daily delivered dose during intensive care stay
  * Filter life span

SECONDARY OUTCOMES:
patient survival | 28-day and 90-day patient survivals

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078
- [Derived] Stucker F, Ponte B, Tataw J, Martin PY, Wozniak H, Pugin J, Saudan P. Efficacy and safety of citrate-based anticoagulation compared to heparin in patients with acute kidney injury requiring continuous renal replacement therapy: a randomized controlled trial. Crit Care. 2015 Mar 18;19(1):91. doi: 10.1186/s13054-015-0822-z. PMID 25881975